CLINICAL TRIAL: NCT04196764
Title: Estudio Observacional Del Seguimiento Prospectivo de la evolución Del Dolor en Pacientes Con Artrosis Primaria de Rodilla Tratados Con Pronolis® HD
Brief Title: Prospective Observational Study of Pain Evolution in Patients With Primary Knee Osteoarthritis Treated With Pronolis® HD
Acronym: NO-DOLOR
Status: Completed | Type: Observational
Sponsor: Procare Health Iberia S.L. (Industry)
Collaborators: Adknoma Health Research (Industry)
Responsible Party: Sponsor
Other Study IDs: NO-DOLOR-2017-01
Record Dates: First submitted 2019-12-11; First posted 2019-12-12 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2019-12

CONDITIONS: Osteo Arthritis Knee

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective observational study of 6 months of follow-up, of national and multicenter scope with medical device with CE marking and according to the usual clinical practice.

In addition, due to the observational design of the clinical investigation, no assignment of the patients will be made to any specific study group, but will be carried out in accordance with the usual clinical practice, not applying any intervention other than the usual one in this type of care practice and always in accordance with current clinical guidelines and recommendations and with the indications authorized in Spain.

Patients will be recruited by specialists and will be followed for 6 months under the conditions of usual clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes and over 18 years.
2. Patients with a previous diagnosis of primary knee osteoarthritis according to ACR criteria and who have a knee x-ray performed during the previous 18 months.
3. Patients who attend a control clinic for primary osteoarthritis of symptomatic knee.
4. Patients with pain equal to or greater than 4 on the VAS scale.
5. Patients who have been prescribed an injection of Pronolis® HD as part of the usual clinical practice.
6. Patients who have given their written informed consent to participate in the clinical investigation.
7. Patients for whom there is a reasonable expectation of follow-up during the development of clinical research.
8. Patients who understand and can complete the questionnaires and do not have cognitive impairment that prevents it.

Exclusion Criteria:

1. Patients with known intolerance to hyaluronic acid.
2. Patients with hypersensitivity to intraarticular injections.
3. Patients who present with infection in the knee joint.
4. Patients presenting with a skin disorder or infection in the area of injection or systemic.
5. Coagulation disorders that contraindicate puncture.
6. Patients who have been prescribed intra-articular injection in both knees.
7. Patients diagnosed with autoimmune rheumatologic diseases or connective diseases.
8. Patients diagnosed with microcrystalline diseases.
9. Patients with traumatic history in the study joint.
10. Patients with a surgical history in the study joint.
11. Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be made up of subjects of legal age diagnosed with primary knee osteoarthritis who have pain equal to or greater than 4 measured by VAS.
  All patients included in this clinical investigation must have been duly informed by the investigator about the investigation procedure and its objectives.
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2017-05-28 (Actual); Primary Completion 2019-02-21 (Actual); Study Completion 2019-10-21 (Actual)

PRIMARY OUTCOMES:
evolution of pain in patients diagnosed with primary knee osteoarthritis 3 months after being treated with hyaluronic acid | 3 months
  3-month baseline change in the domain A score of the WOMAC questionnaire pain will be analyzed to evaluate pain evolution.

SECONDARY OUTCOMES:
evolution of pain in patients diagnosed with primary knee osteoarthritis during the study | 15 days, 1 and 6 months
  Changes in the domain A score of the WOMAC questionnaire pain will be analyzed to evaluate pain evolution.
Pain evolution in motion | 15 days, 1, 3 and 6 months
  Average score of question A1 of the WOMAC questionnaire will be described at each study visit in order to evaluate pain evolution in motion of the affected joint.
stiffness evolution | 15 days, 1, 3 and 6 months
  Average score of domain B of the WOMAC questionnaire will be described at each study visit in order to evaluate the evolution of the stiffness of the affected joint of the patient. In addition, the changes produced between the follow-up visits and the baseline visit will be studied.
evolution of the patient's functional capacity | 15 days, 1, 3 and 6 months
  Average C domain score of the WOMAC questionnaire will be described at each study visit in orde to assess the evolution of the patient's functional capacity. In addition, the changes produced between the follow-up visits and the baseline visit will be studied.
evolution of the patient's quality of life | 3 months
  Average score in the 5 dimensions of the Health Questionnaire EQ-5D-5L (mobility, personal care, usual activities, pain / discomfort, anxiety / depression) at the baseline visit and the 3 month visit in order to evaluate the evolution of the patient's quality of life. In addition, the changes produced between the 3-month visit and the baseline visit will be studied.
satisfaction degree with Pronolis® HD | 15 days, 1, 3 and 6 months
  A likert type scale will be used to assess the patient's satisfaction degree with study treatment in each of the study visits. The evolution of the satisfaction degree (an 5-point Likert Scale) contains 5 items. Higher scores reflected better satisfaction degree
overall clinical impression | 15 days, 1, 3 and 6 months
  For the evaluation of the overall clinical impression of the change by the patient, the ICG-C score will be described in all follow-up visits.
tolerability of treatment with Pronolis® HD | 15 days, 1, 3 and 6 months
  percentage of patients who present adverse effects to the treatment during the observation period will be described in order to evaluate the tolerability of hyaluronic acid treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Calvet J, Khorsandi D, Tio L, Monfort J. Evaluation of a single-shot of a high-density viscoelastic solution of hyaluronic acid in patients with symptomatic primary knee osteoarthritis: the no-dolor study. BMC Musculoskelet Disord. 2022 May 11;23(1):442. doi: 10.1186/s12891-022-05383-w. PMID 35546401